CLINICAL TRIAL: NCT05048862
Title: The Neuroimage Study of the Neuromuscular Disorders.
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201705058RIND
Record Dates: First submitted 2021-08-23; First posted 2021-09-17 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Neuromuscular Diseases
Keywords: neuromuscular disorder; neuromuscular ultrasonography; skin biopsy; muscle biopsy; nerve biopsy; magnetic resonance imaging; electrophysiological study
MeSH Terms: conditions — Neuromuscular Diseases | interventions — Ultrasonography; Nerve Conduction Studies; Genome; Transcriptome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — The DNA, RNA, and protein of the tissues (blood, muscle, nerve and skin) were retrieved and stored in the -80°C refrigerator. The next generation sequencing (whole exon sequencing or whole genome sequencing) and RNA-seq would be performed by NGS & Microarray Core lab in National Taiwan University or another professional team. The protein analysis would be performed by the Proteomics & Protein Function Core Lab in National Taiwan University.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Neuromuscular disorder: Patients age at least 20 years, and have been diagnosed as neuromuscular disorders by the neurologist. Patients who are unable to read the questionnaire, fail to accept all the examinations, and refuse to provide inform consent are excluded from this study.
  Interventions: Diagnostic Test: Neuromuscular ultrasound; Diagnostic Test: Muscle MRI; Diagnostic Test: Nerve conduction studies and autonomic function tests; Diagnostic Test: Quantitative sensory test; Diagnostic Test: Skin biopsy; Diagnostic Test: Muscle and nerve biopsy; Diagnostic Test: Genomics, transcriptome, and proteomics; Diagnostic Test: Laboratory of blood chemical substances, metals and endocrine profiles; Diagnostic Test: Contact heat evoked potentials; Diagnostic Test: Nerve excitability study; Diagnostic Test: Transcranial magnetic stimulation (TMS); Diagnostic Test: fMRI acquisition and image analysis
- Normal group: The normal group (age at least 20 years) who had no neurological symptoms or signs were also recruited. The neurological examination performed by the board neurologist must be normal in the normal group.
  Interventions: Diagnostic Test: Neuromuscular ultrasound; Diagnostic Test: Muscle MRI; Diagnostic Test: Nerve conduction studies and autonomic function tests; Diagnostic Test: Quantitative sensory test; Diagnostic Test: Genomics, transcriptome, and proteomics; Diagnostic Test: Laboratory of blood chemical substances, metals and endocrine profiles; Diagnostic Test: Contact heat evoked potentials; Diagnostic Test: Nerve excitability study; Diagnostic Test: Transcranial magnetic stimulation (TMS); Diagnostic Test: fMRI acquisition and image analysis

INTERVENTIONS:
Diagnostic Test: Neuromuscular ultrasound — Ultrasound will be performed with the Affiniti 70 (Philips Medical Instruments, Bothell, WA). all patients following standardized methods of our hospital. All the patient would be checked the skin surface temperature before the ultrasound examination. The image would be exported from the echo machine as DICOM format.
  Other Names: Sonography
Diagnostic Test: Muscle MRI — Muscle MRI will be performed on a 3-T MR machine (Trio; Siemens, Erlangen, Germany). Each subject will lie in a supine position comfortably, supplied with ear plugs. A high resolution T1 weighted scan and Short-T1 Inversion Recovery series (STIR) of the four limbs muscle were obtained in axial and coronal plane. MR spectroscopy in interested muscle was also sampled to evaluate the composition of fat, water, lactate, and other studied molecules.
Diagnostic Test: Nerve conduction studies and autonomic function tests — Nerve conduction study will be performed with a Nicolet Viking IV Electromyographer (Madison, WI) in all patients following standardized methods recommended by the Consensus Development Conference on Standardized Measures in Diabetic Neuropathy. Studied nerves include sural, peroneal, tibial, median and ulnar (motor and sensory) nerves.Autonomic functions will be assessed by the SSR and RRIV with established protocol by using Nicolet Viking IV Electromyographer (Madison, WI).
Diagnostic Test: Quantitative sensory test — Quantative sensory test will be performed with a Thermal Sensory Analyzer and Vibratory Sensory Analyzer (Medoc Advanced Medical System, Minneapolis, MN). The procedure is the same as previously described 25. Briefly, the machine delivers to the patient a stimulus of constant intensity which is pre-set by the algorithm. By adjusting the intensity of stimulus (increase or decrease the intensity by a fixed ratio) according to the response of the subject (i.e. whether the subject perceives the stimulus or not), sensory thresholds of the warm, cold and vibratory modalities will be measured.
Diagnostic Test: Skin biopsy — A skin specimen of 3 mm in diameter will be taken with a biopsy punch from the lateral side of the distal leg under 2% lidocaine local anaesthesia 26. No suturing is required, and the wounds are covered with a piece of gauze. Wound healing takes 7~10 days, similar to a typical abrasion wound. Informed consent will be obtained from each patient before the skin biopsy. The intraepidermal nerve fiber density and sweat gland nerve innervation will be examined.
  Groups: Neuromuscular disorder
Diagnostic Test: Muscle and nerve biopsy — Two muscle specimens with 5 x 5 x 5 mm were collected in an open muscle biopsy or needle biopsy at studied muscles under 2% lidocaine local anaesthesia. The wound was about 2-3 cm long, and suture was required. Would healing usually takes 10-14 days. First specimen was undergoing snap freezing fixation in a longitudinal axis perpendicular to the cork with the liquid nitrogen and isopentane. The second specimen was divided into two equiponderous tissues, and one was freezed in liquid nitrogen for DNA and protein analysis. The another one was treated with RNAlater solution in 4°C overnight for RNA analysis. Sural nerve biopsies or superficial peroneal nerve were obtained from a standard site posterior to the lateral malleolus under local anesthesia. The nerves were then fixed in 5% glutaraldehyde in 0.1 M phosphate buffer (PB) at 4 °C overnight. All samples were stored in the -80°C refrigerator for further analysis.
  Groups: Neuromuscular disorder
Diagnostic Test: Genomics, transcriptome, and proteomics — The DNA, RNA, and protein of the tissues (blood, muscle, nerve and skin) were retrieved and stored in the -80°C refrigerator. The next generation sequencing (whole exon sequencing or whole genome sequencing) and RNA-seq would be performed by NGS & Microarray Core lab in National Taiwan University or another professional team. The protein analysis would be performed by the Proteomics & Protein Function Core Lab in National Taiwan University.
Diagnostic Test: Laboratory of blood chemical substances, metals and endocrine profiles — The methods of the measurement will follow the standards set by Department of Laboratory Medicine of National Taiwan University Hospital.
Diagnostic Test: Contact heat evoked potentials — A contact heat evoked potential stimulator (Medoc, Ramat Yishai, Israel) will be used for delivering heat stimulation. Stimuli will be delivered repeatedly to the same stimulation site and the inter-stimulus interval will be randomly set to around 18~22 s. CHEP will be recorded using a Nicolet Bravo evoked potential system (Nicolet Biomedical, Madison, WI). The recording electrode was placed at the Cz and P3 of international 10-20 system. The impendence of all recording electrodes was kept below 3 kΩ. The evoked potentials were filtered with a bandpass filter at 0.1~30 Hz. Recording was triggered by the onset of each stimulus, and the sweep time was 1500 ms.
Diagnostic Test: Nerve excitability study — Nerve excitability studies will be undertaken on the median, tibial, peroneal and sural nerves as per previously detailed protocols. Skin temperature will be monitored at the site of stimulation and was maintained at >32°C. Stimulation and recording will be controlled by automated computerized system (QTRAC; Institute of Neurology, London, U.K.) and the stimulus current will be administered using an isolated linear bipolar constant-current stimulator (DS5; Digitimer, Welwyn Garden City, U.K.). Responses will be amplified (ICP511 AC amplifier, Grass Technologies, West Warwick, USA) with electronic noise removed (Hum Bug 50/60 Hz Noise Eliminator, Quest Scientific Instruments, North Vancouver, Canada).
Diagnostic Test: Transcranial magnetic stimulation (TMS) — In simple rTMS protocols, individual stimuli are spaced apart by identical interstimulus intervals (ISI). The stimulation protocol was in accordance with published safety recommendations. The patterned rTMS protocols included (1) Theta burst stimulation, (2) Repetitive paired-pulse TMS. All the above stimulation protocols or paradigms will follow the international guideline of the use of TMS in clinical practice and research (Rossi et al., 2009; Fitzgerald and Daskalakis, 2012; Groppa et al., 2012; Steeves et al., 2012).
Diagnostic Test: fMRI acquisition and image analysis — fMRI will be performed on a 3-T MR machine (Trio; Siemens, Erlangen, Germany). Each subject's head will be positioned comfortably inside a receive-only 8-channel birdcage head coil, supplied with ear plugs, heavily padded and secured with a strap across the forehead in order to minimize head motion. All data will be processed using SPM2 (Wellcome Department of Cognitive Neurology, London UK) 36 implemented on MATLAB (Mathworks Inc. Sherborn, MA).

SUMMARY:
The neuromuscular disorders could be briefly divided to neuropathy, myopathy, motor neuron disease, and neuromuscular junction disorder. In the past, the evaluation of the neuromuscular disorders depended on several ways (ex. electrodiagnostic studies and biopsy) to evaluate the pathophysiology and the pathological change. However, due to the issue of resolution, few image studies were available to evaluate the structure for clinical practice. With the growing techniques, there are two ways to see the nerve and muscle in vivo, the magnetic resonance imaging (MRI) and the ultrasonography. The availability of the machine, the high cost, inability to change the position for dynamic views of the nerves, and the relative invasion considering the large energy penetrating the patient might limit the clinical use of MRI. The nerve ultrasonography is a safe and easily available technique. The development of high-frequency transducers has led to an improvement in the resolution of ultrasonography and enables the exploration of peripheral nerve and muscle structural changes. In additional to evaluate the morphological changes, ultrasonography has been used extensively for the vessel status assessment through duplex ultrasound. In present study, we will apply variable approaches, including to muscle, nerve, and skin biopsy, electrophysiological study, quantitative sensory testing, autonomic functional tests, pain evoked potentials, MRI, and ultrasonography to integrally investigate the different aspects of neuromuscular disorders. The results of the study will provide integrated insights of (1) the neurophysiology of nerve and vessels and (2) pathogenesis of different neuromuscular disorders.

DETAILED DESCRIPTION:
This is a prospective observational study which will be performed in both the inpatient and outpatient setting of National Taiwan University Hospital. Patients age at least 20 years, and have been diagnosed as neuromuscular disorders by the neurologist. Patients who are unable to read the questionnaire, fail to accept all the examinations, and refuse to provide inform consent are excluded from this study. The normal group (age at least 20 years) who had no neurological symptoms or signs were also recruited. The neurological examination performed by the board neurologist must be normal in the normal group.

Different interventions were performed periodically to see the serial change. The interval between the interventions is within 1 month and there is no new symptoms or any events.

ELIGIBILITY:
Inclusion Criteria (Neuromuscular group):

* been diagnosed as neuromuscular disorders by the neurologist
* at least 20-year-old

Inclusion Criteria (Normal group):

* no past history of neurological disorders.
* The neurological examination performed by the board neurologist must be normal
* at least 20-year-old

Exclusion Criteria (Neuromuscular and normal group):

* Patients who are unable to read the questionnaire, fail to accept all the examinations, and refuse to provide inform consent

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients age at least 20 years, and have been diagnosed as neuromuscular disorders by the neurologist. Patients who are unable to read the questionnaire, fail to accept all the examinations, and refuse to provide inform consent are excluded from this study. The normal group (age at least 20 years) who had no neurological symptoms or signs were also recruited. The neurological examination performed by the board neurologist must be normal in the normal group.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2031-08-01 (Estimated); Study Completion 2031-08-01 (Estimated)

PRIMARY OUTCOMES:
Lean muscle volume and fat fraction in MRI | up to 10 years
  Change from Baseline to serial follow-up MRI with the interval of 2 years.
Muscle thickness and echogenecity in ultrasound | up to 10 years
  Change from Baseline to serial follow-up ultrasound with the interval of 2 years.

SECONDARY OUTCOMES:
Natural History | up to 10 years
  To delineate the natural history of different neuromuscular disorders.
Separate disease functional score | up to 10 years
  Separate disease functional scores were: (1) Revised Amyotrophic Lateral Sclerosis Functional Rating Scale (ALSFRS-R) in ALS. The values are 0-48. A lower score indicates a worse outcome. (2) Neuropathy Impairment Score (NIS) and Nerve Disability Score (NDS) in polyneuropathy. The values are 0-244 in NIS and 0-172 in NDS. A higher score indicates a worse outcome in both scores. (3) Medical Research Council Sum-Score (MRC-SS) in myopathy. The values are 0-60. A lower score indicates a worse outcome. (4) MG Activities of Daily Living (MG-ADL) and the Quantitative Myasthenia Gravis (QMG) Test in myasthenia gravis. The values are 0-24 in MG-ADL and 0-72 in QMG. A higher score indicates a worse outcome in both scores.

CONTACTS AND LOCATIONS:
Overall Officials: Hsueh-Wen Hsueh, MD, MMS, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan Univeristy Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Garg N, Park SB, Vucic S, Yiannikas C, Spies J, Howells J, Huynh W, Matamala JM, Krishnan AV, Pollard JD, Cornblath DR, Reilly MM, Kiernan MC. Differentiating lower motor neuron syndromes. J Neurol Neurosurg Psychiatry. 2017 Jun;88(6):474-483. doi: 10.1136/jnnp-2016-313526. Epub 2016 Dec 21. PMID 28003344
- [Background] Pham M, Baumer P, Meinck HM, Schiefer J, Weiler M, Bendszus M, Kele H. Anterior interosseous nerve syndrome: fascicular motor lesions of median nerve trunk. Neurology. 2014 Feb 18;82(7):598-606. doi: 10.1212/WNL.0000000000000128. Epub 2014 Jan 10. PMID 24415574
- [Background] Stewart JD. Magnificent MRI and fascinating selective nerve fascicle damage. Neurology. 2014 Feb 18;82(7):554-5. doi: 10.1212/WNL.0000000000000132. Epub 2014 Jan 10. No abstract available. PMID 24415569
- [Background] Baumer P, Kele H, Xia A, Weiler M, Schwarz D, Bendszus M, Pham M. Posterior interosseous neuropathy: Supinator syndrome vs fascicular radial neuropathy. Neurology. 2016 Nov 1;87(18):1884-1891. doi: 10.1212/WNL.0000000000003287. Epub 2016 Sep 28. PMID 27683851
- [Background] Yoo Y, Kim SJ, Oh J. Postpartum sciatic neuropathy: Segmental fractional anisotropy analysis to disclose neurapraxia. Neurology. 2016 Aug 30;87(9):954-5. doi: 10.1212/WNL.0000000000003051. No abstract available. PMID 27572428
- [Background] Diaz-Manera J, Llauger J, Gallardo E, Illa I. Muscle MRI in muscular dystrophies. Acta Myol. 2015 Dec;34(2-3):95-108. PMID 27199536
- [Background] Huang YN, Chuang HJ, Hsueh HW, Huang HC, Lee NC, Chao CC, Huang PH, Lee YC, Lin KP, Yang CC, Hsieh ST. A case of GNE myopathy mimicking hereditary motor neuropathy. Eur J Neurol. 2020 Nov;27(11):2389-2391. doi: 10.1111/ene.14489. PMID 32860282
- [Background] Buchberger W, Judmaier W, Birbamer G, Lener M, Schmidauer C. Carpal tunnel syndrome: diagnosis with high-resolution sonography. AJR Am J Roentgenol. 1992 Oct;159(4):793-8. doi: 10.2214/ajr.159.4.1529845.
- [Background] Chuang HJ, Hsiao MY, Wu CH, Ozcakar L. Dynamic Ultrasound Imaging for Ulnar Nerve Subluxation and Snapping Triceps Syndrome. Am J Phys Med Rehabil. 2016 Jul;95(7):e113-4. doi: 10.1097/PHM.0000000000000466. No abstract available. PMID 26945221
- [Background] Wu CH, Chang KV, Ozcakar L, Hsiao MY, Hung CY, Shyu SG, Wang TG, Chen WS. Sonographic tracking of the upper limb peripheral nerves: a pictorial essay and video demonstration. Am J Phys Med Rehabil. 2015 Sep;94(9):740-7. doi: 10.1097/PHM.0000000000000344. PMID 26135374
- [Background] Kim BJ, Date ES, Lee SH, Yoon JS, Hur SY, Kim SJ. Distance measure error induced by displacement of the ulnar nerve when the elbow is flexed. Arch Phys Med Rehabil. 2005 Apr;86(4):809-12. doi: 10.1016/j.apmr.2004.08.006. PMID 15827936
- [Background] Chang KV, Lin CP, Hung CY, Ozcakar L, Wang TG, Chen WS. Sonographic Nerve Tracking in the Cervical Region: A Pictorial Essay and Video Demonstration. Am J Phys Med Rehabil. 2016 Nov;95(11):862-870. doi: 10.1097/PHM.0000000000000557. PMID 27362696
- [Background] Hung CY, Hsiao MY, Ozcakar L, Chang KV, Wu CH, Wang TG, Chen WS. Sonographic Tracking of the Lower Limb Peripheral Nerves: A Pictorial Essay and Video Demonstration. Am J Phys Med Rehabil. 2016 Sep;95(9):698-708. doi: 10.1097/PHM.0000000000000463. PMID 26945217
- [Background] Gallardo E, Noto Y, Simon NG. Ultrasound in the diagnosis of peripheral neuropathy: structure meets function in the neuromuscular clinic. J Neurol Neurosurg Psychiatry. 2015 Oct;86(10):1066-74. doi: 10.1136/jnnp-2014-309599. Epub 2015 Feb 4. PMID 25653385
- [Background] Ebadi H, Siddiqui H, Ebadi S, Ngo M, Breiner A, Bril V. Peripheral Nerve Ultrasound in Small Fiber Polyneuropathy. Ultrasound Med Biol. 2015 Nov;41(11):2820-6. doi: 10.1016/j.ultrasmedbio.2015.06.011. Epub 2015 Aug 28. PMID 26318562
- [Background] Gonzalez NL, Hobson-Webb LD. Neuromuscular ultrasound in clinical practice: A review. Clin Neurophysiol Pract. 2019 Jul 12;4:148-163. doi: 10.1016/j.cnp.2019.04.006. eCollection 2019. PMID 31886438
- [Background] Adler RS, Garolfalo G, Paget S, Kagen L. Muscle sonography in six patients with hereditary inclusion body myopathy. Skeletal Radiol. 2008 Jan;37(1):43-8. doi: 10.1007/s00256-007-0367-6. Epub 2007 Oct 26. PMID 17962939
- [Background] Evans KD, Roll SC, Volz KR, Freimer M. Relationship between intraneural vascular flow measured with sonography and carpal tunnel syndrome diagnosis based on electrodiagnostic testing. J Ultrasound Med. 2012 May;31(5):729-36. doi: 10.7863/jum.2012.31.5.729. PMID 22535720
- [Background] Vanderschueren GA, Meys VE, Beekman R. Doppler sonography for the diagnosis of carpal tunnel syndrome: a critical review. Muscle Nerve. 2014 Aug;50(2):159-63. doi: 10.1002/mus.24241. Epub 2014 Jul 14. PMID 24633597
- [Background] Carandang MAE, Takamatsu N, Nodera H, Mori A, Mimura N, Okada N, Kinoshita H, Kuzuya A, Urushitani M, Takahashi R, Izumi Y, Kaji R. Velocity of intraneural blood flow is increased in inflammatory neuropathies: sonographic observation. J Neurol Neurosurg Psychiatry. 2017 May;88(5):455-457. doi: 10.1136/jnnp-2016-314547. Epub 2016 Nov 25. No abstract available. PMID 27888186
- [Background] Angus-Leppan H, Burke D. The function of large and small nerve fibers in renal failure. Muscle Nerve. 1992 Mar;15(3):288-94. doi: 10.1002/mus.880150306. PMID 1313545
- [Background] Chao CC, Tsai LK, Chiou YH, Tseng MT, Hsieh ST, Chang SC, Chang YC. Peripheral nerve disease in SARS:: report of a case. Neurology. 2003 Dec 23;61(12):1820-1. doi: 10.1212/01.wnl.0000099171.26943.d0. No abstract available. PMID 14694063
- [Background] Gutrecht JA. Sympathetic skin response. J Clin Neurophysiol. 1994 Sep;11(5):519-24. doi: 10.1097/00004691-199409000-00006. PMID 7844242
- [Background] Stalberg EV, Nogues MA. Automatic analysis of heart rate variation: I. Method and reference values in healthy controls. Muscle Nerve. 1989 Dec;12(12):993-1000. doi: 10.1002/mus.880121207. PMID 2622473
- [Background] Pan CL, Lin YH, Lin WM, Tai TY, Hsieh ST. Degeneration of nociceptive nerve terminals in human peripheral neuropathy. Neuroreport. 2001 Mar 26;12(4):787-92. doi: 10.1097/00001756-200103260-00034. PMID 11277584
- [Background] Chien HF, Tseng TJ, Lin WM, Yang CC, Chang YC, Chen RC, Hsieh ST. Quantitative pathology of cutaneous nerve terminal degeneration in the human skin. Acta Neuropathol. 2001 Nov;102(5):455-61. doi: 10.1007/s004010100397. PMID 11699558
- [Background] Hsieh ST, Lin WM. Modulation of keratinocyte proliferation by skin innervation. J Invest Dermatol. 1999 Oct;113(4):579-86. doi: 10.1046/j.1523-1747.1999.00737.x. PMID 10504444
- [Background] Pan CL, Tseng TJ, Lin YH, Chiang MC, Lin WM, Hsieh ST. Cutaneous innervation in Guillain-Barre syndrome: pathology and clinical correlations. Brain. 2003 Feb;126(Pt 2):386-97. doi: 10.1093/brain/awg039. PMID 12538405
- [Background] Granovsky Y, Matre D, Sokolik A, Lorenz J, Casey KL. Thermoreceptive innervation of human glabrous and hairy skin: a contact heat evoked potential analysis. Pain. 2005 Jun;115(3):238-247. doi: 10.1016/j.pain.2005.02.017. Epub 2005 Apr 18. PMID 15911150
- [Background] Valeriani M, Le Pera D, Niddam D, Chen AC, Arendt-Nielsen L. Dipolar modelling of the scalp evoked potentials to painful contact heat stimulation of the human skin. Neurosci Lett. 2002 Jan 18;318(1):44-8. doi: 10.1016/s0304-3940(01)02466-1. PMID 11786221
- [Background] Chen AC, Niddam DM, Arendt-Nielsen L. Contact heat evoked potentials as a valid means to study nociceptive pathways in human subjects. Neurosci Lett. 2001 Dec;316(2):79-82. doi: 10.1016/s0304-3940(01)02374-6. PMID 11742720
- [Background] Chao CC, Hsieh ST, Chiu MJ, Tseng MT, Chang YC. Effects of aging on contact heat-evoked potentials: the physiological assessment of thermal perception. Muscle Nerve. 2007 Jul;36(1):30-8. doi: 10.1002/mus.20815. PMID 17503497
- [Background] Chen AC, Niddam DM, Crawford HJ, Oostenveld R, Arendt-Nielsen L. Spatial summation of pain processing in the human brain as assessed by cerebral event related potentials. Neurosci Lett. 2002 Aug 9;328(2):190-4. doi: 10.1016/s0304-3940(02)00512-8. PMID 12133585
- [Background] Kiernan MC, Lin CS, Andersen KV, Murray NM, Bostock H. Clinical evaluation of excitability measures in sensory nerve. Muscle Nerve. 2001 Jul;24(7):883-92. doi: 10.1002/mus.1085. PMID 11410915
- [Background] Bostock H, Cikurel K, Burke D. Threshold tracking techniques in the study of human peripheral nerve. Muscle Nerve. 1998 Feb;21(2):137-58. doi: 10.1002/(sici)1097-4598(199802)21:23.0.co;2-c. PMID 9466589
- [Background] Friston KJ, Holmes AP, Poline JB, Grasby PJ, Williams SC, Frackowiak RS, Turner R. Analysis of fMRI time-series revisited. Neuroimage. 1995 Mar;2(1):45-53. doi: 10.1006/nimg.1995.1007. PMID 9343589
- [Background] Collins DL, Neelin P, Peters TM, Evans AC. Automatic 3D intersubject registration of MR volumetric data in standardized Talairach space. J Comput Assist Tomogr. 1994 Mar-Apr;18(2):192-205. PMID 8126267
- [Background] Buchel C, Holmes AP, Rees G, Friston KJ. Characterizing stimulus-response functions using nonlinear regressors in parametric fMRI experiments. Neuroimage. 1998 Aug;8(2):140-8. doi: 10.1006/nimg.1998.0351. PMID 9740757